CLINICAL TRIAL: NCT00544440
Title: An Observational Study of Continuous Oral Dosing of an Irreversible CYP17 Inhibitor, Abiraterone Acetate (CB7630), in Castration-Resistant Prostate Cancer Patients Evaluating Androgens and Steroid Metabolites in Bone Marrow Plasma
Brief Title: An Observational Study of Continuous Oral Dosing of Abiraterone Acetate in Castration-Resistant Prostate Cancer Patients Evaluating Androgens and Steroid Metabolites in Bone Marrow Plasma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR016906; COU-AA-BMA (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2007-10-15; First posted 2007-10-16 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Prostate Neoplasms
Keywords: Prostate neoplasms; Prostate cancer; Castration-resistant prostate cancer; Abiraterone acetate; CB7630; Prednisone; Testosterone; Bone marrow
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abiraterone acetate plus prednisone (Experimental): Patients will be treated orally with abiraterone acetate 1000 mg daily and prednisone 5 mg twice a day until clinical disease progression.
  Interventions: Drug: Abiraterone acetate; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone acetate — Abiraterone 1000 mg (4 x 250 mg tablets) taken orally once daily
Drug: Prednisone — Prednisone 5 mg tablet taken orally twice daily

SUMMARY:
The purpose of this study is to investigate the effect of abiraterone acetate on levels of androgens and steroid metabolites in bone marrow plasma of patients with metastatic castration-resistant prostate cancer (CRPC).

DETAILED DESCRIPTION:
This is a single-center, open-label (identity of assigned study drug will be known) study investigating the effect of abiraterone acetate on levels of testosterone and dihydrotestosterone (DHT) in bone marrow plasma of patients with metastatic CRPC and evaluating the difference in bone marrow androgen levels between patients with and without serum prostate specific antigen (PSA) decline. Approximately 60 medically or surgically castrated male patients with metastatic CRPC will be enrolled. The study will consist of screening, treatment, and follow-up periods. Patients will be treated orally (by mouth) with abiraterone acetate 1000 mg daily and prednisone 5 mg twice a day until clinical disease progression. Follow-up will continue until the patient dies, is lost to follow-up or withdraws informed consent. Bone marrow aspirates will be collected at Week 1 (predose), Week 9, and the final study visit. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the prostate
* Eastern Cooperative Oncology Group (ECOG) performance status <=2 (Karnofsky Performance Status >=50%)
* Serum testosterone levels <50ng/ml
* Ongoing gonadal androgen deprivation therapy with luteinizing hormone-releasing hormone (LHRH) analogues or orchiectomy (patients, who have not had an orchiectomy, must be maintained on effective LHRH analogue therapy for the duration of the study)
* Progression of disease despite androgen ablation (either documented osseous or soft tissue metastatic disease progression or by prostate specific antigen [PSA] criteria progression)
* Progressive disease is defined by PSA evidence (PSA level of at least 5 ng/ml which has risen on at least 2 successive occasions, at least 2 weeks apart)
* Presence of metastatic bone disease
* Discontinue diethylstilbestrol or steroids treatment for >=4 weeks and for antiandrogens >6 weeks
* Antiandrogen withdrawal: patients who are receiving an antiandrogen as part of primary androgen ablation must demonstrate disease progression following discontinuation of antiandrogen (disease progression after antiandrogen withdrawal is defined as 2 consecutive rising PSA values, obtained at least 2 weeks apart, or documented osseous or soft tissue progression)
* For patients receiving flutamide, at least one of the PSA values must be obtained 4 weeks or more after flutamide discontinuation
* For patients receiving bicalutamide or nilutamide, at least one of the PSA values must be obtained 6 weeks or more after antiandrogen discontinuation
* Adequate adrenal function
* Laboratory values within protocol -defined parameters
* No evidence of chronic or acute disseminated intravascular coagulation or bleeding tendency and no angina at rest
* Agrees to protocol-defined use of effective contraception

Exclusion Criteria:

* Histologic variants other than adenocarcinoma in the primary tumor
* More then 2 different prior chemotherapeutic regimens for metastatic prostate cancer
* Abnormal liver function
* Therapy with other hormonal therapy, including any dose of megestrol acetate (Megace), Ketoconazole, finasteride (Proscar), dutasteride (Avodart) any herbal product known to decrease PSA levels (eg, Saw Palmetto and PC-SPES), or any systemic corticosteroid within 4 weeks prior to first dose of study drug
* Active infection or intercurrent illness that are not controlled
* Unstable angina, myocardial infarction within the previous 6 months, or use of ongoing maintenance therapy for life-threatening ventricular arrhythmia, uncontrolled hypertension, New York Heart Association (NYHA) Class III or IV congestive heart failure
* Prior radiation therapy completed <4 weeks or single fraction of palliative radiotherapy within 14 days prior to first dose of study drug
* Any currently active second malignancy, other than non-melanoma skin cancer
* Active psychiatric illnesses/social situations that would limit compliance with protocol requirements
* Active or uncontrolled autoimmune disease that may require corticosteroid therapy during study
* Severely compromised immunological state, including being positive for the human immunodeficiency virus (HIV)
* Acute or chronic hepatitis B or C
* Initiation of bisphosphonate therapy within 4 weeks prior to first dose of study drug
* Long QT syndrome or bundle branch block or hemiblock or other history of life-threatening arrhythmia (unless the patient has been effectively treated for it and is considered stable)
* Known brain metastasis
* History of pituitary or adrenal dysfunction
* History of gastrointestinal disorders (medical disorders or extensive surgery) which may interfere with the absorption of the study drug
* Prior therapy with abiraterone acetate
* Any acute toxicities due to prior chemotherapy and/or radiotherapy that have not resolved to a NCI CTCAE (version 3) grade of <=1
* Condition or situation which, in the investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-10; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Houston, Texas, United States

REFERENCES:
- See also: NATIONAL CANCER INSTITUTE — http://www.cancer.gov
- See also: NATIONAL INSTITUTE OF HEALTH — http://www.nlm.nih.gov/medlineplus/prostatecancer.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Abiraterone Acetate: Patients were treated orally with abiraterone acetate 1000 mg daily and prednisone 5 mg twice a day until clinical disease progression.
Period: Overall Study
Arm/Group | Abiraterone Acetate
Started | 57
Completed | 0
Not Completed | 57
Not completed — Other | 1
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 2
Not completed — Subject Non-compliance | 1
Not completed — Progressive Disease | 47
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.1 (8.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 57

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Detectable Bone Marrow Testosterone Level (>1 Picograms/Mililiter)
Time Frame: Baseline (predose Week 1 Day 1) and Week 8
Population: Bone marrow aspirates were collected at baseline (predose Week 1 Day 1) in 49 participants and in 44 participants at Week 8.
Measure: Number; unit: Number of Participants
Groups:
- Abiraterone Acetate: Participants were treated orally with abiraterone acetate 1000 mg daily and prednisone 5 mg twice a day until clinical disease progression.
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 49
Number of Participants
  Baseline (predose Week 1 Day 1) (n=49) | 0
  Week 8 (n=44) | 0

2. Primary Outcome: Number of Participants With Detectable Bone Marrow Dihydrotestosterone (DHT) Level (>9 Picograms/Mililiter)
Time Frame: Baseline (predose Week 1 Day 1) and Week 8
Population: as for outcome 1
Measure: Number; unit: Number of Participants
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 49
Number of Participants
  Baseline (predose Week 1 Day 1) (n=49) | 2
  Week 8 (n=44) | 2

3. Primary Outcome: Difference in Bone Marrow Testosterone Levels Between Participants With and Without Serum Prostate Specific Antigen Decline
Time Frame: Week 8
Population: Since there were too few participants with any detectable bone marrow testosterone, this analysis was not performed.
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Change in Markers of Bone Metabolism
Time Frame: Week 8
Population: Data was reported in individual participant listings but not summarized due to statistical constraints.
Arm/Group | Abiraterone Acetate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Abiraterone Acetate
Serious Adverse Events (participants affected / at risk) | 29/57
Other Adverse Events (participants affected / at risk) | 56/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=57)
Anaemia (Blood and lymphatic system disorders) | 3
Coagulopathy (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Acute myocardial infarction (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Disease progression (General disorders) | 3
Fatigue (General disorders) | 3
Pyrexia (General disorders) | 1
Catheter related infection (Infections and infestations) | 1
Infection (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood bicarbonate decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Weight decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Paraplegia (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 2
Confusional state (Psychiatric disorders) | 1
Mood altered (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Urinary tract obstruction (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 3
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone Acetate (N=57)
Anaemia (Blood and lymphatic system disorders) | 30
Leukopenia (Blood and lymphatic system disorders) | 5
Lymphopenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Constipation (Gastrointestinal disorders) | 15
Diarrhoea (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 3
Flatulence (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 36
Oedema peripheral (General disorders) | 20
Pyrexia (General disorders) | 5
Hyperbilirubinaemia (Hepatobiliary disorders) | 10
Urinary tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 12
Alanine aminotransferase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 15
Blood albumin decreased (Investigations) | 3
Blood alkaline phosphatase increased (Investigations) | 36
Blood bilirubin increased (Investigations) | 6
Blood calcium decreased (Investigations) | 3
Blood cholesterol increased (Investigations) | 9
Blood creatinine increased (Investigations) | 11
Blood glucose increased (Investigations) | 3
Blood triglycerides increased (Investigations) | 8
Platelet count decreased (Investigations) | 4
White blood cell count decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 11
Hypercholesterolaemia (Metabolism and nutrition disorders) | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 47
Hyperkalaemia (Metabolism and nutrition disorders) | 5
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 16
Hypoalbuminaemia (Metabolism and nutrition disorders) | 26
Hypocalcaemia (Metabolism and nutrition disorders) | 11
Hypoglycaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 20
Hypomagnesaemia (Metabolism and nutrition disorders) | 12
Hyponatraemia (Metabolism and nutrition disorders) | 12
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 22
Back pain (Musculoskeletal and connective tissue disorders) | 23
Bone pain (Musculoskeletal and connective tissue disorders) | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 8
Neuropathy peripheral (Nervous system disorders) | 5
Peripheral motor neuropathy (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 5
Pollakiuria (Renal and urinary disorders) | 4
Pelvic pain (Reproductive system and breast disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10
Dry skin (Skin and subcutaneous tissue disorders) | 9
Hypertension (Vascular disorders) | 24
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.